CLINICAL TRIAL: NCT01192061
Title: Autonomic Nervous System Activity, Peripheral Microcirculation and Retrobulbar Hemodynamics in Normal Tension Glaucoma Patients.
Brief Title: Autonomic Nervous System Activity and Normal Tension Glaucoma
Acronym: ANS
Status: Completed | Type: Observational
Sponsor: Military Institute od Medicine National Research Institute (Other)
Collaborators: Polish Academy of Sciences (Other); Indiana University School of Medicine (Other); Medical University of Warsaw (Other)
Responsible Party: Joanna Wierzbowska, MD, Military Medical Instutute, Department of Ophthalmology
Other Study IDs: N N402 165637
Record Dates: First submitted 2010-08-30; First posted 2010-08-31 (Estimated); Last update posted 2011-01-25 (Estimated); Status verified 2011-01

CONDITIONS: Normal Tension Glaucoma
Keywords: autonomic nervous system; heart rate variability; blood pressure variability; retrobulbar hemodynamics; vascular dysregulation
MeSH Terms: conditions — Low Tension Glaucoma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Normal tension glaucoma group
- Control group

SUMMARY:
Evidence has accumulated that systemic and ocular mechanisms, responsible for regulating blood flow in the area of the optic disc, such as reduced ocular perfusion pressure, abnormal autoregulation and vascular dysregulation may be involved in the pathogenesis of normal tension glaucoma (NTG). Defective cardiovascular neuroregulation has been advocated as a possible one of the main systemic contributing factors in the etiology of NTG. Based on the results of previous studies, the hypothesis has been posed that patients with NTG have an impaired diurnal heart rate variability (HRV) or high activity of the sympathetic component of autonomic nervous system (ANS) and endothelial dysfunction. Impaired balance of ANS, resulting in increased demand for oxygen in the tissues and subsequent low threshold of hypoxia in all organs (including the eye) can be an important link in the pathogenetic pathway of NTG, making the optic nerve more sensitive to small and short-term changes in perfusion pressure and prone to damage even under a statistically "normal" intraocular pressure (IOP).

The aim of this study is to evaluate the activity and characteristics of the following systems: the central ANS (through a 24-hour analysis of heart rate variability and blood pressure), peripheral vascular system (through the analysis of the post-occlusive hyperemia reaction within the distal part of left upper limb) and the local retrobulbar circulation as measured by color Doppler imaging (CDI) in patients with NTG and healthy volunteers. The correlations between all above systems, as well as between them and the structural and functional parameters of the optic nerve, and the retina in both groups will be also analyzed.

DETAILED DESCRIPTION:
Fifty patients with NTG and 50 age and gender-matched control subjects will be recruited. All patients will be underwent eye examination (medical history, best corrected visual acuity, slit-lamp and stereo optic disc evaluation, Goldmann applanation tonometry, central corneal thickness measurement , Humphrey central 24-2 threshold perimetry test and optical coherence tomography of the optic nerve head, retinal nerve fibre layer and macula. CDI examination of the retrobulbar vessels will be performed. 24-hour ambulatory electrocardiogram and blood pressure monitoring will be performed simultaneously. Time- and frequency-domain measures of HRV will be calculated. BP will be measured in 20 minutes intervals during the day and 30 minutes intervals at night. The occlusive provocative test and finger hyperemia will be assessed by two-channels laser-Doppler flowmeter.

ELIGIBILITY:
Inclusion Criteria:

NTG group

* both gender
* early to moderate NTG
* without significant cardiac or pulmonary conditions. Glaucoma is diagnosed on the basis of a glaucomatous appearance of the optic disc (cup-to-disc ratio greater than 0.6 or an interocular cup-to-disc ratio asymmetry greater than or equal to 0.2, and at least one of the following abnormalities: thinning of the rim, notching, nerve fiber layer defects, or peripapillary atrophy), correlating with visual field defects in two consecutive central 24-2 program of Humphrey threshold perimetry, according to the European Glaucoma Society (EGS) diagnostic criteria (abnormal glaucoma hemifield test or cluster of three non-edge contiguous points at the <5% level on the pattern deviation plot with at least one point at the <1% level, with < 25% fixation losses and false positives and false negatives responses). Early and moderately glaucomatous loss is defined according to the Hodapp et al. classification, based on the Mean Defect (MD) index of visual fields less than - 6 dB (decibels) and - 12 dB but more than -6 dB, respectively, and on the basis of a vertical cup/disc ratio less than 0.8.

Control group

* both gender
* age and gender-matched
* without glaucoma
* without significant cardiac or pulmonary conditions.

Exclusion Criteria:

* ocular hypertension
* primary open angle glaucoma (high pressure glaucoma, IOP>21mmHg)
* secondary open angle glaucoma
* angle closure glaucoma
* history of eye surgery
* history of eye trauma
* myopia above -6.0 diopters (D)
* corneal dystrophies
* uncontrolled arterial hypertension
* atrial fibrillation
* atrial flutter
* pacemaker
* history of cardiac arrest
* vasovagal syndrome
* diabetes mellitus
* primary damage to the autonomic nervous system
* Shy-Drager syndrome
* encephalomyelitis, multiple sclerosis
* brain and spinal cord tumors
* renal failure
* carotid sinus hypersensitivity syndrome carotid sinus
* carotid artery stenosis
* pregnancy
* breast-feeding

Min Age: 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: NTG group: out-patient clinic of the Ophthalmology Department of the Military Medical Institute (MMI), control group: hospital stuff, family and friends of hospital stuff and patients
Sampling Method: Non-Probability Sample
Enrollment: 97 (Actual)
Dates: Start 2010-02; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Time and spectral-domain measures of heart rate variability | baseline
  standard deviation of normal to normal RR intervals (SDNN), standard deviation of normal to normal RR intervals index (SD SD), root mean square of succesive differences (RMS-SD), percentage of normal to normal RR interval, greater than 50 ms (pNN50), low-frequency component (LF), high frequency component (HF), LF/HF) ratio

SECONDARY OUTCOMES:
retrobulbar hemodynamic parameters of ophthalmic (OA), central retinal (CRA) and short ciliary posterior arteries (SCPA) | baseline
  peak systolic velocity (PSV) of OA, CRA and SPCA, end diastolic velocity (EDV) of OA, CRA and SPCA, resistance index (RI) of OA, CRA and SPCA
measures of blood pressure (BP) diurnal variability | baseline
  standard devation of of the average systolic BP (SD SBP24), diastolic BP (SD DBP24) and mean BP (SD MBP24) during the whole day, standard devation of of the average systolic BP (SD SBPd), diastolic BP (SD DBPd) and mean BP (SD MBPd) during the day and standard devation of of the average systolic BP (SD SBPn), diastolic BP (SD DBPn) and mean BP (SD MBPn) at night.
parameters of postocclusive hyperemia response | baseline
  biological zero (BZ) (mean flow signal during occlusion), maximum hyperemia response (MAX) (maximum flow signal of post-occlusive hyperemia response), time of recovery (TR) (time from the end of occlusion until the moment when flow signal returns to the rest values), time to peak-flow (TM) (time from the moment of the end of occlusion until the moment of maximum hyperemic response), and half time of hyperemia (TH) (time from the moment of the end of occlusion until the moment when flow signal reaching the maximum value will fall by half)
optical coherence tomography parameters of optic nerve head | baseline
  disc area (DA), cup area (CA), rim area (RA), cup/disc area ratio (CDR), cup/disc horizontal ratio (CDHR), cup/disc vertical ratio (CDVR)
optical coherence tomography parameters of the retinal nerve fibre layer (RNFL) | baseline
  mean RNFL thickness (RNFL M), mean inferior RNFL thickness (RNFL I), mean superior RNFL thickness (RNFL S), mean temporal RNFL thickness (RNFL T), mean nasal RNFL thickness (RNFL N).
optical coherence tomography parameters of macula | baseline
  minimum macula thickness (TF MIN), mean macula thickness (TF M), mean inferior interior macula thickness (IIM), mean superior interior macula thickness (SIM), mean nasal interior macula thickness (NIM), mean temperal interior macula thickness (TIM), mean inferior outer macula thickness (IOM), mean superior outer macula thickness (SOM), mean nasal outer macula thickness (NOM), mean temporal outer macula thickness (TOM), volume foveola (VF) and volume macula (VM).
Parameters of visual field examination | baseline
  mean defect (MD), pattern standard deviation (PSD)

CONTACTS AND LOCATIONS:
Overall Officials: Joanna Wierzbowska, MD, PhD, Principal Investigator — Military Medical Institute, Department of Ophthalmology, 128 Szaserow Str. 04-141 Warsaw, Poland
Locations (1):
- Military Medical Institute, Warsaw, Poland

REFERENCES:
- [Background] Wierzbowska J, Wierzbowski R, Stankiewicz A, Robaszkiewicz J. [Autonomic nervous system and primary open angle glaucoma--pathogenetic and clinical correlations]. Klin Oczna. 2009;111(1-3):75-9. Polish. PMID 19517852
- [Background] Brown CM, Dutsch M, Michelson G, Neundorfer B, Hilz MJ. Impaired cardiovascular responses to baroreflex stimulation in open-angle and normal-pressure glaucoma. Clin Sci (Lond). 2002 Jun;102(6):623-30. PMID 12049615
- [Background] Riccadonna M, Covi G, Pancera P, Presciuttini B, Babighian S, Perfetti S, Bonomi L, Lechi A. Autonomic system activity and 24-hour blood pressure variations in subjects with normal- and high-tension glaucoma. J Glaucoma. 2003 Apr;12(2):156-63. doi: 10.1097/00061198-200304000-00011. PMID 12671471
- [Background] Kashiwagi K, Tsumura T, Ishii H, Ijiri H, Tamura K, Tsukahara S. Circadian rhythm of autonomic nervous function in patients with normal-tension glaucoma compared with normal subjects using ambulatory electrocardiography. J Glaucoma. 2000 Jun;9(3):239-46. doi: 10.1097/00061198-200006000-00007. PMID 10877375